CLINICAL TRIAL: NCT01417416
Title: Changes in the Permeability of the Blood Brain Barrier and Intestinal Barrier in Humans During Conditions of Stress and Immune Activation: in Vivo Studies
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: C/08/236; DSOCL08210 (Other Grant/Funding Number: DSTA Singapore)
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2009-02

CONDITIONS: Combat Training Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- with combat training stress
- without combat training stress

SUMMARY:
The relevance of BBB and IB permeability changes as a major precipitating cause for cognitive and digestive dysfunction in the military stress setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male troops (aged 18-50 yrs) scheduled to be engaged in a protracted multi-day stressful field exercises.

Exclusion Criteria:

* Significantly systemic disease, including cardiovascular, psychiatric, neurological (including polyneuropathies) and endocrine disease including diabetes mellitus.
* No written informed consent obtained from subject.

Ages: 18 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: Healthy male troops during combat training
Sampling Method: Probability Sample